CLINICAL TRIAL: NCT05657132
Title: Antibacterial Effect of New Herbal Paste Used as an Intracanal Medication in Necrotic Primary Molars, a Randomized Control Trial
Brief Title: Antibacterial Effect of New Herbal Paste Used as an Intracanal Medication
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nahda University (Other)
Responsible Party: Principal Investigator, GHada Abdelwahab Ahmed, Associate Professor of Pediatric Dentistry, Nahda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 050622
Record Dates: First submitted 2022-12-10; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Infection Primary
Keywords: infected primary molars, metapaste, herbal paste

STUDY DESIGN:
Intervention Model Description: randomized control trial
Who Masked: Participant
Masking Description: blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Costus paste (Experimental): Costus paste used as an intracanal medication for decreasing the number of enterococcus faecalis present in the necrotic root of the primary molar
  Interventions: Drug: herbal intracanal medication paste
- metapaste (Active Comparator): metapaste used as an intracanal medication for decreasing the number of enterococcus faecalis present in the necrotic root of the primary molar
  Interventions: Drug: Meta paste

INTERVENTIONS:
Drug: herbal intracanal medication paste — study the effect of costus herbal paste on enterococcus faecalis bacteria
  Other Names: herbal paste
  Arms: Costus paste
Drug: Meta paste — compare the effect of Costus paste with meta paste in reducing the number of enterococcus faecalis
  Other Names: control paste
  Arms: metapaste

SUMMARY:
studying the antibacterial effect of Cosuts paste as an intracanal medication against Enterococcus faecalis that present in necrotic primary teeth

DETAILED DESCRIPTION:
The children were randomly divided into two groups (I, II) Group I (N=12): using Costus-based paste as an intracanal medicament. Group II (N= 12): Calcium hydroxide iodoform paste (Metapex) as an intracanal medicament.

Procedure:

Access opening was started. then a swab was taken from the distal root canal with a dry paper point and transferred to a sterile test tube. The canals were filled with an intracanal medication according to the patient group. In group I, the canals was filled with a previously prepared Costus-based paste for one week, and In Group II, the canals were filled with Meta paste for one week. After 1 week, the paste was washed away from the canals then another swab was taken from the distal canal by a dry paper point as done before preoperatively.

The 2 swabs were transferred within 2 hours to the lab for bacterial culture and detection of enterococcus faecalis count.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically and radiologically diagnosed infected primary teeth in their mandibular arch.
* Teeth should be deeply carious, with a history of spontaneous pain and carious exposures with necrotic pulp was also be selected
* radiographic evidence of adequate alveolar bone support, and absence of internal or external resorption.
* tooth must be restorable.

Exclusion Criteria:

* vital tooth
* Non restorable teeth

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Bacterial count | 1 weak
  Colony forming unit

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Salem, Ph.D, Principal Investigator — associate professor of Pediatric Dentistry
Locations (1):
- NUB University, Cairo, Bani Suif, Egypt

IPD SHARING:
Plan to Share IPD: No
not to share IPD until publication